CLINICAL TRIAL: NCT04291508
Title: Acetaminophen and Ascorbate in Sepsis: Targeted Therapy to Enhance Recovery
Acronym: ASTER
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Boyd Taylor Thompson, PETAL CCC Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PETAL04ASTER
Record Dates: First submitted 2020-02-27; First posted 2020-03-02 (Actual); Results first posted 2024-09-27 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Acute Respiratory Distress Syndrome; Critical Illness; Respiratory Failure; Sepsis
Keywords: ARDS; Acetaminophen; Vitamin C; Sepsis
MeSH Terms: conditions — Respiratory Distress Syndrome; Critical Illness; Respiratory Insufficiency; Sepsis | interventions — Glucose

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to at a ratio of 2:1 active versus placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Vitamin C or Vitamin C-placebo will be refrigerated. Acetaminophen or acetaminophen-placebo will be stored at room temperature and the volume will be reduced for patients less than 50 kg. Investigators will be informed of which of the two placebo controlled groups the patient was randomized to.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- IV Acetaminophen-Active (Active Comparator): Patients randomized to the Acetaminophen arm will receive Acetaminophen at the dose of 1 gram (or 15 mg/kg if actual body weight < 50kg) in 100 ml 5% dextrose in water every 6 hours intravenously for 5 days (20 doses).
  Interventions: Drug: Intravenous Acetaminophen (room temperature)
- IV Vitamin C-Active (Active Comparator): Patients randomized to the Vitamin C arm will receive Vitamin C at the dose of 50 mg/kg in 100 ml 5% dextrose in water every 6 hours intravenously for 5 days (20 doses). Note: This arm is now closed.
  Interventions: Drug: Intravenous Vitamin C (refrigerated)
- Acetaminophen-Placebo (Placebo Comparator): Patients randomized to placebo will receive an identical-appearing intravenous infusion of 100 ml of 5% dextrose in water every 6 hours for 5 days (20 doses).
  Interventions: Drug: 5% Dextrose (room temperature)
- Vitamin C-Placebo (Placebo Comparator): Patients randomized to placebo will receive an identical-appearing intravenous infusion of 100 ml of 5% dextrose in water every 6 hours for 5 days (20 doses). Note: This arm is now closed.
  Interventions: Drug: 5% Dextrose refrigerated

INTERVENTIONS:
Drug: Intravenous Acetaminophen (room temperature) — Acetaminophen given intravenously at the dose of 1 gram (or 15 mg/kg if patient weighs < 50 kg) every six hours for 5 days (20 doses)
  Arms: IV Acetaminophen-Active
Drug: Intravenous Vitamin C (refrigerated) — Vitamin C given intravenously at the dose of 50 mg/kg every six hours for 5 days (20 doses)
  Other Names: Ascor
  Arms: IV Vitamin C-Active
Drug: 5% Dextrose (room temperature) — Placebo (identical appearing room temperature 5% dextrose solution) infused every six hours for 5 days (20 doses)
  Arms: Acetaminophen-Placebo
Drug: 5% Dextrose refrigerated — Placebo (identical appearing refrigerated 5% dextrose solution) infused every six hours for 5 days (20 doses)
  Arms: Vitamin C-Placebo

SUMMARY:
Prospective multi-center phase 2b randomized placebo-controlled double-blinded interventional platform trial of two different pharmacologic therapies (intravenous Vitamin C or intravenous Acetaminophen) for patients with sepsis-induced hypotension or respiratory failure.

DETAILED DESCRIPTION:
Hypothesis 1A: Acetaminophen (APAP) or Vitamin C infusion will increase the days alive and free of organ support to day 28.

Hypothesis 1B: APAP or Vitamin C will have a favorable effect on other secondary outcomes including pulmonary and non-pulmonary organ dysfunction and biomarkers of inflammation and endothelial injury

The investigators plan to carry out two multi-center phase 2b randomized double-blinded placebo-controlled trials of two different pharmacologic therapies within a single platform trial.

1. One trial will assess the efficacy of Acetaminophen (1 gram intravenously every 6 hours) for 120 hours in patients with sepsis who have evidence of either hemodynamic or respiratory organ failure.
2. A second trial will assess the efficacy of Vitamin C (50 mg/kg every 6 hours) infused intravenously for 120 hours in patients with sepsis who have evidence of either hemodynamic or respiratory organ failure.

A total of 900 participants who meet all of the inclusion criteria and none of the exclusion criteria, were planned be randomized in a 2:1:2:1 fashion (APAP-Active: APAP-Placebo: Vit C-Active: Vit C-Placebo). The APAP and Vitamin C trials were planned to be resulted separately. With the closure of the Vitamin C arm in June 2022; the study proceeded with the APAP and Placebo arms with a 1:1 randomization scheme. The total sample size for the APAP trial was 447 participants (227 in the active arm and 220 in the placebo arm). The total sample size for the Vitamin C trial was 79 (40 in the active arm and 39 in the placebo arm). The total combined number in the 4 arms of the ASTER trial was 526 (227 APAP active, 220 APAP placebo, 40 Vit C active, 39 Vit C placebo), although a total of only 487 patients were actually randomized (this is due to the 39 pooled placebo patients that appear in both trials).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Sepsis defined as:

   1. Clinical evidence of a known or suspected infection and orders written to administer antibiotics AND
   2. Hypotension as defined by the need for any vasopressor (and 1 liter of fluid already administered intravenously for resuscitation) OR respiratory failure defined by mechanical ventilation, BIPAP or CPAP at any level, or greater than or equal to 6 liters/minute of supplemental oxygen (criterion b must be met at time of enrollment)
3. Admitted to a study site ICU (or intent for the patient to be admitted to a study site ICU) within 36 hours of presentation to the ED or admitted to the study site ICU within 36 hours of presentation to any acute care hospital

Exclusion Criteria:

1. No consent/inability to obtain consent from the participant or a legally authorized representative
2. Patient unable to be randomized within 36 hours of presentation to the ED or within 36 hours of presentation to any acute care hospital
3. Diagnosis of cirrhosis by medical chart review
4. Liver transplant recipient
5. AST or ALT greater than five times upper limit of normal
6. Diagnosis of ongoing chronic alcohol use disorder/abuse by chart review; if medical record unclear, use Appendix F
7. Clinical diagnosis of diabetic ketoacidosis or other condition such as profound hypoglycemia that requires hourly blood glucose monitoring (applicable to the 4 arm (Vitamin C/placebo vs. Acetaminophen/placebo) phase of the trial)
8. Hypersensitivity to Acetaminophen or Vitamin C
9. Patient, surrogate or physician not committed to full support (Exception: a patient will not be excluded if he/she would receive all supportive care except for attempts at resuscitation from cardiac arrest)
10. Home assisted ventilation (via tracheotomy or noninvasive) except for CPAP/BIPAP used only for sleep-disordered breathing
11. Chronic dialysis
12. Current active kidney stone (applicable to the 4 arm (Vitamin C/placebo vs. Acetaminophen/placebo) phase of the trial)
13. Multiple (>1) episodes of prior kidney stones, known history of oxalate kidney stones, or history of oxalate nephropathy. (applicable to the 4 arm (Vitamin C/placebo vs. Acetaminophen/placebo) phase of the trial)
14. Kidney transplant recipient (applicable to the 4 arm (Vitamin C/placebo vs. Acetaminophen/placebo) phase of the trial)
15. Use of home oxygen >3L/minute via nasal cannula for chronic cardiopulmonary disease
16. Moribund patient not expected to survive 24 hours
17. Underlying malignancy or other condition with estimated life expectancy of less than 1 month
18. Pregnant woman, woman of childbearing potential without a documented negative urine or serum pregnancy test during the current hospitalization, or woman who is breast feeding
19. Prisoner
20. Treating team unwilling to enroll because of intended use of Acetaminophen or Vitamin C
21. Treating team unwilling to use plasma (as opposed to point of care testing) for glucose monitoring (applicable to the 4 arm (Vitamin C/placebo vs. Acetaminophen/placebo) phase of the trial).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 488 (Actual)
Dates: Start 2021-10-13 (Actual); Primary Completion 2023-04-27 (Actual); Study Completion 2023-07-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boyd Taylor Thompson, MD, Principal Investigator — Massachusetts General Hospital
Locations (41):
- United States (41):
  - University of Alabama Medical Center, Birmingham, Alabama
  - University of Arizona, Tucson, Arizona
  - UCSF Fresno, Fresno, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - UC Davis Medical Center, Sacramento, California
  - UCSF Medical Center, San Francisco, California
  - Stanford University, Stanford, California
  - University of Colorado Hospital, Aurora, Colorado
  - Denver Health Medical Center, Denver, Colorado
  - University Medical Center, New Orleans, Louisiana
  - Maine Medical Center, Portland, Maine
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - University of Michigan Medical Center, Ann Arbor, Michigan
  - Henry Ford Medical Center, Detroit, Michigan
  - Fairview Southdale Hospital, Edina, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Mt. Sinai Hospital, New York, New York
  - Montefiore Medical Center-Weiler, The Bronx, New York
  - Montefiore Medical Center-Moses, The Bronx, New York
  - Carolinas Medical Center, Charlotte, North Carolina
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Wexner Medical Center, Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Temple University Hospital, Philadelphia, Pennsylvania
  - UPMC Presbyterian/Mercy/Shadyside/Magee, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas Health Science Center, Houston, Texas
  - Intermountain Medical Center, Murray, Utah
  - University of Utah Hospital, Salt Lake City, Utah
  - University of Virginia Health System, Charlottesville, Virginia
  - Sentara/EVMS, Norfolk, Virginia
  - VCU Medical Center, Richmond, Virginia
  - Harborview Medical Center, Seattle, Washington
  - Swedish Hospital First Hill, Seattle, Washington

REFERENCES:
- [Derived] Ware LB, Files DC, Fowler A, Aboodi MS, Aggarwal NR, Brower RG, Chang SY, Douglas IS, Fields S, Foulkes AS, Ginde AA, Harris ES, Hendey GW, Hite RD, Huang W, Lai P, Liu KD, Thompson BT, Matthay MA; National Heart, Lung, and Blood Institute Prevention and Early Treatment of Acute Lung Injury Clinical Trials Network. Acetaminophen for Prevention and Treatment of Organ Dysfunction in Critically Ill Patients With Sepsis: The ASTER Randomized Clinical Trial. JAMA. 2024 Aug 6;332(5):390-400. doi: 10.1001/jama.2024.8772. PMID 38762798
- See also: Website for the PETAL Network — http://petalnet.org

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There were 488 participants randomized overall. 228 to APAP, 199 to matching APAP placebo, 40 to Vit C, 21 to matching Vit C placebo. Thirty-nine patients appear in both placebo arms in our published results (these were pooled placebos). Clinical Trials.gov does not allow reporting pooled placebo patients twice in each of these two studies. Therefore, the results reported herein don't mirror our published results which were reported per protocol and as specified in our SAP.
Groups:
- Acetaminophen-Placebo: Patients randomized to APAP matching placebo (initially 2:1, subsequently 1:1 after the Vitamin C arm stopped) will receive an identical-appearing intravenous infusion of 100 ml of 5% dextrose in water every 6 hours for 5 days (20 doses).
  5% Dextrose (room temperature): Placebo (identical appearing room temperature 5% dextrose solution) infused every six hours for 5 days (20 doses).
- Vitamin C-Placebo: Patients randomized to matching Vitamin C placebo (2:1) will receive an identical-appearing intravenous infusion of 100 ml of 5% dextrose in water every 6 hours for 5 days (20 doses). Note: This arm is now closed.
  5% Dextrose refrigerated: Placebo (identical appearing refrigerated 5% dextrose solution) infused every six hours for 5 days (20 doses)
Period: Overall Study
Arm/Group | IV Acetaminophen-Active | IV Vitamin C-Active | Acetaminophen-Placebo | Vitamin C-Placebo
Started | 228 | 40 | 199 | 21
Completed | 223 | 40 | 197 | 21
Not Completed | 5 | 0 | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 0
Not completed — lost to follow up | 4 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: There were 487 participants randomized. For baseline variables that were missing, the measure analysis population differs from the baseline analysis population. For these variables, a footnote identifies the reason for the discrepancy.
Groups:
- Total: Total of all reporting groups
Arm/Group | IV Acetaminophen-Active | IV Vitamin C-Active | Acetaminophen-Placebo | Vitamin C-Placebo | Total
Number analyzed (Participants) | 227 | 40 | 199 | 21 | 487
Age, Continuous [Mean (Standard Deviation); unit: years] — Total column is reported for the 486 patients analyzed. Population: Data for age missing for one patient in the APAP placebo arm; as a result the Total column reflects 486 patients total.
  years
    number analyzed (Participants) | 227 | 40 | 198 | 21 | 486
    (all) | 63.9 (15.9) | 62.4 (17.0) | 63.8 (14.7) | 67.6 (16.4) | 63.9 (15.5)
Age, Customized [Count of Participants; unit: Participants] — Age > 75 years Population: Measure Analysis Population Description: Data for age missing for one patient in the APAP placebo arm; as a result the Total column reflects 486 patients total.
  Participants
    Yes: number analyzed (Participants) | 227 | 40 | 198 | 21 | 486
    Yes | 57 | 10 | 47 | 8 | 122
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 112 | 21 | 102 | 12 | 247
  Male | 115 | 19 | 97 | 9 | 240
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 31 | 3 | 24 | 4 | 62
  Not Hispanic or Latino | 191 | 37 | 170 | 16 | 414
  Unknown or Not Reported | 5 | 0 | 5 | 1 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 0 | 0 | 2
  Asian | 6 | 2 | 12 | 0 | 20
  Native Hawaiian or Other Pacific Islander | 4 | 1 | 3 | 0 | 8
  Black or African American | 45 | 10 | 30 | 2 | 87
  White | 153 | 25 | 131 | 17 | 326
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 17 | 2 | 23 | 2 | 44
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 227 | 40 | 199 | 21 | 487
Baseline total SOFA score (no-GCS) [Mean (Standard Deviation); unit: Units on a scale] — Reported for 487 patients randomized.Higher SOFA score=worse outcome. ASTER clinically sig organ failure: SOFA score >/=2 points higher than baseline. Total score range: 0(min)-24(max) Score: Coag(platelets x10³/µL: 0:>150; 1:</=150; 2:</=100; 3:</=50; 4:</=20. Liver(bilirubin, mg/dL): 0:<1.2; 1: 1.2-1.9; 3: 2.0-5.9; 3: 6.0-11.9; 4:>11.9. Cardio(hypotension): 0:none; 1: MAP <70 mmHg; 2: Dop</=5 or dob (any dose); 3:dop>5, epi</=0.1, or norepi</=0.1; 4: Dop>15, epi>0.1, or norepi>0.1. Renal(Cr, mg/dL or urine output,ml/d): 0:<1.2; 1: 1.2-1.9; 3: 2.0-3.4; 3: 3.5-4.9 or <500; 4:>4.9 or <200.
  Units on a scale | 5.5 (2.5) | 5.2 (2.3) | 5.3 (2.5) | 4.8 (2.4) | 5.3 (2.5)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — Reported for the 486 patients analyzed. Population: BMI is missing in one patient in the APAP placebo arm resulting in only 198 patients with this baseline variable; as a result the Total column reflects 486 patients total.
  kg/m^2
    number analyzed (Participants) | 227 | 40 | 198 | 21 | 486
    (all) | 29.3 (10.2) | 33.9 (17.3) | 29.1 (9.6) | 27.5 (7.4) | 29.5 (10.7)
Vasopressors at baseline no. (%) [Count of Participants; unit: Participants] | 174 | 30 | 152 | 14 | 370
Assisted ventilation at baseline, no. (%) [Count of Participants; unit: Participants] — Population: Baseline assisted ventilation data missing for one patient in the APAP active arm and one patient in the APAP placebo arm.
  Participants
    number analyzed (Participants) | 226 | 40 | 198 | 21 | 485
    (all) | 99 | 17 | 81 | 5 | 202
HFNO at baseline no.(%) [Count of Participants; unit: Participants] — Population: Data for baseline HFNO missing for one patient in the APAP active arm and one patient in the APAP placebo arm.
  Participants
    number analyzed (Participants) | 226 | 40 | 198 | 21 | 485
    (all) | 33 | 6 | 33 | 6 | 78
ARDS at baseline no. (%) [Count of Participants; unit: Participants] — Population: Data for baseline ARDS missing for one patient in the APAP active arm and one patient in the APAP placebo arm.
  Participants
    number analyzed (Participants) | 226 | 40 | 198 | 21 | 485
    (all) | 41 | 10 | 28 | 2 | 81
Time from inclusion to randomization (hour), median (q1-q3) [Median (Inter-Quartile Range); unit: hours] — Total column is reported for the 479 patients we had this data point for. Population: Data missing on time to randomization for 3 patients in the APAP active arm and 5 patients in the APAP placebo arm; as a result the Total column reflects 479 patients total.
  hours
    number analyzed (Participants) | 224 | 40 | 194 | 21 | 479
    (all) | 9.6 [2.9 to 19.0] | 13.2 [4.7 to 19.1] | 9.2 [2.4 to 19.1] | 12.9 [7.4 to 21.5] | 9.8 [2.9 to 19.1]
Screening hospital location no. (%) [Count of Participants; unit: Participants]
  Intensive care unit | 128 | 16 | 123 | 13 | 280
  Emergency department | 95 | 24 | 74 | 8 | 201
  Floor | 2 | 0 | 0 | 0 | 2
  Other | 2 | 0 | 1 | 0 | 3
  stepdown/intermediate unit | 0 | 0 | 1 | 0 | 1
Site of infection no. (%) [Count of Participants; unit: Participants]
  Pneumonia | 100 | 17 | 85 | 11 | 213
  Urinary tract infection | 37 | 8 | 47 | 5 | 97
  Intra-abdominal infection | 24 | 4 | 18 | 1 | 47
  Skin or soft-tissue infection | 17 | 3 | 14 | 2 | 36
  Flu/other virus confirmed by testing | 8 | 1 | 3 | 0 | 12
  Central nervous system infection | 3 | 2 | 4 | 0 | 9
  Endocarditis or endovascular infection | 1 | 1 | 1 | 0 | 3
  Vascular catheter-related infection | 0 | 1 | 1 | 1 | 3
  Other source of infection | 15 | 1 | 6 | 0 | 22
  Unknown to providers | 22 | 2 | 20 | 1 | 45
COVID-19 status in 3 weeks prior to admission no. (%) [Count of Participants; unit: Participants]
  Positive test within 3 weeks prior to admission | 17 | 6 | 18 | 4 | 45
  Negative (only negative tests with 3 weeks prior to admission) | 163 | 28 | 154 | 16 | 361
  Unknown | 47 | 6 | 27 | 1 | 81
Baseline creatinine (mg/dL) [Mean (Standard Deviation); unit: mg/dL] — Total column is reported for the 487 patients randomized.
  mg/dL | 1.6 (1.3) | 1.8 (1.6) | 1.7 (1.3) | 1.4 (1.0) | 1.6 (1.3)
Baseline outpatient creatinine in 365 days prior to admission (mg/dL) [Mean (Standard Deviation); unit: mg/dL] — Total column is reported for the 368 patients who had this lab value available. Population: Numbers in analyzed rows differs from overall because baseline outpatient creatinine was not available for all randomized patients; as a result the Total column reflects 368 patients total.
  mg/dL
    number analyzed (Participants) | 164 | 29 | 157 | 18 | 368
    (all) | 1.1 (0.8) | 1.1 (1.0) | 1.3 (1.1) | 0.9 (0.5) | 1.2 (0.9)
Baseline AST (U/L) [Mean (Standard Deviation); unit: U/L] — Total column is reported for the 487 patients randomized.
  U/L | 45.5 (35.0) | 46.9 (35.9) | 40.4 (37.2) | 45.3 (27.1) | 43.5 (35.7)
Baseline ALT (U/L) [Mean (Standard Deviation); unit: U/L] — Total column is reported for the 487 patients randomized.
  U/L | 30.9 (26.6) | 32.5 (23.6) | 31.0 (34.2) | 35.7 (36.2) | 31.3 (30.1)
Baseline bilirubin (mg/dL) [Mean (Standard Deviation); unit: mg/dL] — Total column is reported for the 483 patients with baseline bilirubin available.. Population: Number analyzed in row differs from overall because we collected clinically available bilirubin and bilirubin values were not available for all randomized patients; as a result the Total column reflects 483 patients total.
  mg/dL
    number analyzed (Participants) | 225 | 40 | 197 | 21 | 483
    (all) | 0.9 (0.9) | 0.8 (0.5) | 0.9 (1.0) | 1.1 (2.1) | 0.9 (1.0)
Baseline platelets (×1000/mm³) [Mean (Standard Deviation); unit: (cells*1000/mm^3)] — Total column is reported for the 486 patients analyzed. Population: Baseline platelets was not available for one patient in the APAP active arm resulting in only 226 patients analyzed in that column; as a result the Total column reflects 486 patients total.
  (cells*1000/mm^3)
    number analyzed (Participants) | 226 | 40 | 199 | 21 | 486
    (all) | 218.9 (125.9) | 208.9 (104.2) | 225.3 (135.5) | 180.7 (107.6) | 219.0 (127.6)
Baseline Plasma cell-free hemoglobin (mg/dL) [Mean (Standard Deviation); unit: mg/dL] — Total column is reported for the 469 patients with Baseline Plasma cell-free hemoglobin available. Population: Baseline Plasma cell-free hemoglobin was missing in 7 APAP active patients and 8 APAP placebo patients resulting in numbers analyzed being different from overall; as a result the Total column reflects 469 patients total.
  mg/dL
    number analyzed (Participants) | 218 | 39 | 192 | 20 | 469
    (all) | 24.1 (60.3) | 26.6 (31.2) | 18.9 (40.7) | 64.9 (167.7) | 23.9 (60.5)
Baseline Acetaminophen no. (%) [Count of Participants; unit: Participants] | 106 | 27 | 84 | 7 | 224
Baseline plasma cell-free Hemoglobin [Median (Inter-Quartile Range); unit: mg/dL] — Total column is reported for the 469 patients with Baseline Plasma cell-free hemoglobin available. Population: Data was not available for all patients for this baseline variable. As a result the Total column reflects 469 patients total.
  mg/dL
    number analyzed (Participants) | 218 | 39 | 192 | 20 | 469
    (all) | 8.3 [4.4 to 17.0] | 14.2 [6.5 to 27.7] | 8.3 [4.6 to 17.1] | 15.9 [4.4 to 50.4] | 8.6 [4.6 to 19.0]

OUTCOME MEASURES:

1. Primary Outcome: Days Alive and Free of Organ Support to Day 28
Description: Defined as the days alive and free of organ support (dialysis, assisted ventilation, and vasopressors) to day 28. Participants will need to be free of all three components (assisted ventilation, vasopressors, new renal replacement therapy) to qualify for a day alive and free from organ failures. Patients on chronic dialysis will not be scored for the new renal failure free component of this outcome.
Time Frame: 28 days after randomization
Population: Data needed to determine this outcome was missing in 4 patients in the Acetaminophen active arm and 2 patients in the Acetaminophen placebo arm.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | IV Acetaminophen-Active | IV Vitamin C-Active | Acetaminophen-Placebo | Vitamin C-Placebo
Number analyzed (Participants) | 223 | 40 | 197 | 21
days | 20.2 (10.6) | 20.5 (9.5) | 19.7 (10.5) | 18.4 (11.7)
Statistical Analysis 1: Comparison: IV Acetaminophen-Active vs Acetaminophen-Placebo; Test type: Superiority; p = 0.65, t-test, 2 sided; Mean Difference (Final Values) = 0.5, 95% CI 2-sided [-1.6 to 2.5]
Statistical Analysis 2: Comparison: IV Vitamin C-Active vs Vitamin C-Placebo; Test type: Superiority; p = 0.464, t-test, 2 sided; Mean Difference (Final Values) = 2.0, 95% CI 2-sided [-3.5 to 7.6]

2. Primary Outcome: 28-day All Cause Mortality
Description: Vital status at study day 28 regardless of location or cause of death. Patients discharged from the study hospital are followed to day 29 to determine this endpoint.
Time Frame: 28 days after randomization
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | IV Acetaminophen-Active | IV Vitamin C-Active | Acetaminophen-Placebo | Vitamin C-Placebo
Number analyzed (Participants) | 223 | 40 | 197 | 21
Participants | 39 | 6 | 43 | 6
Statistical Analysis 1: Comparison: IV Acetaminophen-Active vs Acetaminophen-Placebo; Test type: Superiority; p = 0.26, Chi-squared; Risk Difference (RD) = -4.3, 95% CI 2-sided [-12.0 to 3.3]
Statistical Analysis 2: Comparison: IV Vitamin C-Active vs Vitamin C-Placebo; Test type: Superiority; p = 0.31, Fisher Exact; Risk Difference (RD) = -13.6, 95% CI 2-sided [-35.8 to 8.7]

3. Primary Outcome: Days Free of Assisted Ventilation to Day 28
Description: The number of days alive and without assisted ventilation (midnight to midnight) in the overall cohort. No penalty for death.
Time Frame: 28 days after randomization
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: days
Arm/Group | IV Acetaminophen-Active | IV Vitamin C-Active | Acetaminophen-Placebo | Vitamin C-Placebo
Number analyzed (Participants) | 223 | 40 | 197 | 21
days | 21.5 (10.2) | 21.6 (9.4) | 20.6 (10.5) | 19.5 (11.7)
Statistical Analysis 1: Comparison: IV Acetaminophen-Active vs Acetaminophen-Placebo; Test type: Superiority; p = 0.35, t-test, 2 sided; Mean Difference (Final Values) = 1.0, 95% CI 2-sided [-1.0 to 2.9]
Statistical Analysis 2: Comparison: IV Vitamin C-Active vs Vitamin C-Placebo; Test type: Superiority; p = 0.45, t-test, 2 sided; Mean Difference (Final Values) = 2.1, 95% CI 2-sided [-3.4 to 7.6]

4. Primary Outcome: Days Free of Renal Replacement Therapy to Day 28 in Overall Cohort
Description: The number of days alive and without renal replacement (RRT) in the overall cohort. If a participant was not on RRT at randomization, received RRT every other day, and stopped RRT before day 28, the number of renal replacement free days is the sum of the days free of RRT prior to dialysis starting and the number of days after dialysis stopped (begins with the first day, midnight to midnight, the participant was free of RRT). No penalty for death.
Time Frame: 28 days after randomization
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: days
Arm/Group | IV Acetaminophen-Active | IV Vitamin C-Active | Acetaminophen-Placebo | Vitamin C-Placebo
Number analyzed (Participants) | 223 | 40 | 197 | 21
days | 23.7 (9.0) | 24.8 (7.8) | 23.9 (8.4) | 20.8 (10.9)
Statistical Analysis 1: Comparison: IV Acetaminophen-Active vs Acetaminophen-Placebo; Test type: Superiority; p = 0.83, t-test, 2 sided; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-1.9 to 1.5]
Statistical Analysis 2: Comparison: IV Vitamin C-Active vs Vitamin C-Placebo; Test type: Superiority; p = 0.10, t-test, 2 sided; Mean Difference (Final Values) = 4.0, 95% CI 2-sided [-0.8 to 8.9]

5. Primary Outcome: Days Free of Vasopressors to Day 28 in Overall Cohort
Description: Days free of vasopressors to day 28 are defined as the number of calendar days (midnight to midnight) between randomization and 28 days later that the patient is alive and did not receive vasopressor therapy.
Time Frame: 28 days after randomization
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: days
Arm/Group | IV Acetaminophen-Active | IV Vitamin C-Active | Acetaminophen-Placebo | Vitamin C-Placebo
Number analyzed (Participants) | 223 | 40 | 197 | 21
days | 22.2 (9.4) | 22.6 (8.6) | 23.9 (8.4) | 19.1 (11.3)
Statistical Analysis 1: Comparison: IV Acetaminophen-Active vs Acetaminophen-Placebo; Test type: Superiority; p = 0.55, t-test, 2 sided; Mean Difference (Final Values) = 0.6, 95% CI 2-sided [-1.2 to 2.4]
Statistical Analysis 2: Comparison: IV Vitamin C-Active vs Vitamin C-Placebo; Test type: Superiority; p = 0.18, t-test, 2 sided; Mean Difference (Final Values) = 3.5, 95% CI 2-sided [-1.6 to 8.7]

6. Secondary Outcome: Ventilator-free Days (VFD)
Description: VFDs depend on both duration of ventilation and mortality through study day 28. In participants who survive 28 days, VFD is defined as 28 minus days of invasive or noninvasive ventilation to day 28. Duration of ventilation is counted from the first study day of assisted breathing through the last day of assisted breathing provided the last day is prior to day 28. Isolated periods of ventilation briefer than 24 hours for surgical procedures and ventilation solely for sleep disordered breathing do not count towards duration of ventilation. In participants who never require assisted breathing, duration of ventilation is zero. Participants who do not survive 28 days will be assigned zero VF
Time Frame: 28 days after randomization
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: days
Arm/Group | IV Acetaminophen-Active | IV Vitamin C-Active | Acetaminophen-Placebo | Vitamin C-Placebo
Number analyzed (Participants) | 223 | 40 | 197 | 21
days | 20.9 (11.0) | 21.3 (10.1) | 19.5 (11.8) | 18.8 (12.7)
Statistical Analysis 1: Comparison: IV Acetaminophen-Active vs Acetaminophen-Placebo; Test type: Superiority; p = 0.21, t-test, 2 sided; Mean Difference (Final Values) = 1.4, 95% CI 2-sided [-0.8 to 3.6]
Statistical Analysis 2: Comparison: IV Vitamin C-Active vs Vitamin C-Placebo; Test type: Superiority; p = 0.40, t-test, 2 sided; Mean Difference (Final Values) = 2.5, 95% CI 2-sided [-3.4 to 8.5]

7. Secondary Outcome: Vasopressor-free Days
Description: Vasopressor free days to day 28 are defined as the number of calendar days between randomization and 28 days later that the patient is alive and without the use of vasopressor therapy. Patients who die prior to day 28 and those who receive vasopressor therapy for the entire first 28 days are assigned zero vasopressor free days.
Time Frame: 28 days after randomization
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: days
Arm/Group | IV Acetaminophen-Active | IV Vitamin C-Active | Acetaminophen-Placebo | Vitamin C-Placebo
Number analyzed (Participants) | 223 | 40 | 197 | 21
days | 21.4 (10.4) | 21.8 (10.0) | 20.2 (11.3) | 18.2 (12.3)
Statistical Analysis 1: Comparison: IV Acetaminophen-Active vs Acetaminophen-Placebo; Test type: Superiority; p = 0.23, t-test, 2 sided; Mean Difference (Final Values) = 1.3, 95% CI 2-sided [-0.8 to 3.4]
Statistical Analysis 2: Comparison: IV Vitamin C-Active vs Vitamin C-Placebo; Test type: Superiority; p = 0.22, t-test, 2 sided; Mean Difference (Final Values) = 3.6, 95% CI 2-sided [-2.2 to 9.4]

8. Secondary Outcome: Renal Replacement-free Days
Description: Renal replacement free days to day 28 are defined as the number of calendar days between randomization and 28 days later that the patient is alive and without renal replacement therapy. We also follow the "last off" method. Patients who died prior to day 28 and those who receive renal replacement therapy for the entire first 28 days are assigned zero renal replacement free days.
Time Frame: 28 days after randomization
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: days
Arm/Group | IV Acetaminophen-Active | IV Vitamin C-Active | Acetaminophen-Placebo | Vitamin C-Placebo
Number analyzed (Participants) | 223 | 40 | 197 | 21
days | 22.4 (11.0) | 23.7 (10.1) | 21.8 (11.6) | 19.1 (12.8)
Statistical Analysis 1: Comparison: IV Acetaminophen-Active vs Acetaminophen-Placebo; Test type: Superiority; p = 0.58, t-test, 2 sided; Mean Difference (Final Values) = 0.6, 95% CI 2-sided [-1.6 to 2.8]
Statistical Analysis 2: Comparison: IV Vitamin C-Active vs Vitamin C-Placebo; Test type: Superiority; p = 0.13, t-test, 2 sided; Mean Difference (Final Values) = 4.5, 95% CI 2-sided [-1.4 to 10.5]

9. Secondary Outcome: 28 Day Hospital Mortality
Description: All deaths occuring in the study hospital until study day 28.
Time Frame: 28 days after randomization
Population: Data needed to determine this outcome was missing in 3 patients in the Acetaminophen active arm and 2 patients in the Acetaminophen placebo arm.
Measure: Count of Participants; unit: Participants
Arm/Group | IV Acetaminophen-Active | IV Vitamin C-Active | Acetaminophen-Placebo | Vitamin C-Placebo
Number analyzed (Participants) | 224 | 40 | 197 | 21
Participants | 37 | 6 | 41 | 6
Statistical Analysis 1: Comparison: IV Acetaminophen-Active vs Acetaminophen-Placebo; Test type: Superiority; p = 0.26, Chi-squared; Risk Difference (RD) = -4.3, 95% CI 2-sided [-11.8 to 3.2]
Statistical Analysis 2: Comparison: IV Vitamin C-Active vs Vitamin C-Placebo; Test type: Superiority; p = 0.31, Fisher Exact; Risk Difference (RD) = -13.6, 95% CI 2-sided [-35.8 to 8.7]

10. Secondary Outcome: ICU Free Days
Description: The number of days spent alive out of the ICU to day 28.
Time Frame: 28 days after randomization
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: days
Arm/Group | IV Acetaminophen-Active | IV Vitamin C-Active | Acetaminophen-Placebo | Vitamin C-Placebo
Number analyzed (Participants) | 223 | 40 | 197 | 21
days | 19.3 (9.9) | 18.7 (9.7) | 19.1 (10.0) | 17.9 (12.0)
Statistical Analysis 1: Comparison: IV Acetaminophen-Active vs Acetaminophen-Placebo; Test type: Superiority; p = 0.76, t-test, 2 sided; Mean Difference (Final Values) = 0.3, 95% CI 2-sided [-1.6 to 2.2]
Statistical Analysis 2: Comparison: IV Vitamin C-Active vs Vitamin C-Placebo; Test type: Superiority; p = 0.78, t-test, 2 sided; Mean Difference (Final Values) = 0.8, 95% CI 2-sided [-4.9 to 6.5]

11. Secondary Outcome: Hospital Free Days to Discharge Home
Description: Defined as 28 days minus the number of days from randomization to discharge home. If a patient has not been discharged home prior to study day 28 or dies prior to day 28, hospital free days will be zero. Patients transferred to another hospital or other health care facility will be followed to day 28 to assess this endpoint.
Time Frame: Up to day 28
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: days
Arm/Group | IV Acetaminophen-Active | IV Vitamin C-Active | Acetaminophen-Placebo | Vitamin C-Placebo
Number analyzed (Participants) | 223 | 40 | 196 | 21
days | 11.3 (10.9) | 11.5 (10.0) | 11.5 (10.8) | 7.0 (10.4)
Statistical Analysis 1: Comparison: IV Acetaminophen-Active vs Acetaminophen-Placebo; Test type: Superiority; p = 0.84, t-test, 2 sided; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-2.3 to 1.9]
Statistical Analysis 2: Comparison: IV Vitamin C-Active vs Vitamin C-Placebo; Test type: Superiority; p = 0.10, t-test, 2 sided; Mean Difference (Final Values) = 4.5, 95% CI 2-sided [-0.9 to 10.0]

12. Secondary Outcome: Number of Subjects With Initiation of Assisted Ventilation
Description: Any patient who received assisted ventilation during the study hospitalization to study day 28 days meets this endpoint.
Time Frame: Up to day 28
Measure: Count of Participants; unit: Participants
Arm/Group | IV Acetaminophen-Active | IV Vitamin C-Active | Acetaminophen-Placebo | Vitamin C-Placebo
Number analyzed (Participants) | 125 | 23 | 116 | 16
Participants | 21 | 4 | 21 | 2
Statistical Analysis 1: Comparison: IV Acetaminophen-Active vs Acetaminophen-Placebo; Test type: Superiority; p = 0.79, Chi-squared; Risk Difference (RD) = -1.3, 95% CI 2-sided [-10.9 to 8.3]
Statistical Analysis 2: Comparison: IV Vitamin C-Active vs Vitamin C-Placebo; Test type: Superiority; p = 1.00, Fisher Exact; Risk Difference (RD) = 4.9, 95% CI 2-sided [-17.5 to 27.3]

13. Secondary Outcome: Number of Subjects With Initiation of Renal Replacement Therapy
Description: Patients who receive (new) renal replacement therapy through day 28 will meet this endpoint. Patients with chronic renal replacement therapy initiated prior to the current sepsis illness will not be eligible to meet this endpoint.
Time Frame: Up to day 28
Measure: Count of Participants; unit: Participants
Arm/Group | IV Acetaminophen-Active | IV Vitamin C-Active | Acetaminophen-Placebo | Vitamin C-Placebo
Number analyzed (Participants) | 223 | 40 | 197 | 21
Participants | 22 | 3 | 16 | 2
Statistical Analysis 1: Comparison: IV Acetaminophen-Active vs Acetaminophen-Placebo; Test type: Superiority; p = 0.53, Chi-squared; Risk Difference (RD) = 1.7, 95% CI 2-sided [-3.7 to 7.2]
Statistical Analysis 2: Comparison: IV Vitamin C-Active vs Vitamin C-Placebo; Test type: Superiority; p = 1.00, Fisher Exact; Risk Difference (RD) = -2.0, 95% CI 2-sided [-17.0 to 13.0]

14. Secondary Outcome: Change in Organ-specific Sepsis-related Organ Failure Assessment (SOFA) Scores Between Enrollment and Study Day 7
Description: SOFA score calculated upon enrollment and at day 7 using clinically available data. If a value is not available at baseline, it will be assumed to be normal. Missing values at day 7 assessment were carried forward to the closest known value. GSC was omitted for patients intubated/heavily sedated at either 0 or day 7 when calculating the change in score. Renal dysfunction component was omitted for patients RRT prior to presentation.Higher SOFA score=worse outcome.ASTER clinically significant organ failure:SOFA score 2 or more points higher than baseline.Total score range: 0(min)-24(max) Score:Coag(platelets x10³/µL:0:>150;1:</=150; 2:</=100; 3:</=50; 4:</=20. Liver(bilirubin, mg/dL): 0:<1.2; 1: 1.2-1.9; 3: 2.0-5.9; 3: 6.0-11.9; 4:>11.9. Cardio(hypotension): 0:none; 1: MAP <70 mmHg; 2: Dop</=5 or dob (any dose); 3:dop>5, epi</=0.1, or norepi</=0.1; 4: Dop>15, epi>0.1, or norepi>0.1. Renal(Cr, mg/dL or urine output,ml/d): 0:<1.2; 1: 1.2-1.9; 3: 2.0-3.4; 3: 3.5-4.9 or <500; 4:>4.9 or<200.
Time Frame: Day 0-Day 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IV Acetaminophen-Active | IV Vitamin C-Active | Acetaminophen-Placebo | Vitamin C-Placebo
Number analyzed (Participants) | 148 | 28 | 139 | 14
score on a scale | -3.2 (3.3) | -2.2 (4.6) | -3.0 (3.2) | -2.1 (2.1)
Statistical Analysis 1: Comparison: IV Acetaminophen-Active vs Acetaminophen-Placebo; Test type: Superiority; p = 0.70, t-test, 2 sided; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-0.9 to 0.6]
Statistical Analysis 2: Comparison: IV Vitamin C-Active vs Vitamin C-Placebo; Test type: Superiority; p = 0.96, t-test, 2 sided; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-2.7 to 2.5]

15. Secondary Outcome: Renal Calculi to Day 90
Description: Renal calculi diagnosed between randomization and study day 90 in patients in the Vitamin C-Active/Vitamin C-Placebo group.
Time Frame: Up to day 90
Population: Renal calculi diagnosed between randomization and study day 90 in patients in the Vitamin C-Active/Vitamin C-Placebo group.
Measure: Count of Participants; unit: Participants
Arm/Group | IV Acetaminophen-Active | IV Vitamin C-Active | Acetaminophen-Placebo | Vitamin C-Placebo
Number analyzed (Participants) | 0 | 40 | 0 | 21
Participants | 0 | 1 | 0 | 0
Statistical Analysis 1: Comparison: IV Vitamin C-Active vs Vitamin C-Placebo; Test type: Superiority; p = 1.00, Fisher Exact; Risk Difference (RD) = 2.5, 95% CI 2-sided [-2.3 to 7.3]

16. Secondary Outcome: 90-day All-cause Mortality
Description: Vital status of the patient at day 90 will be determined using any of the following methods: medical record review, phone calls to patient, proxy or healthcare facility, review of obituaries, or information from the Centers for Disease Control and Prevention's National Death Index (NDI).
Time Frame: 90 days after randomization
Measure: Count of Participants; unit: Participants
Arm/Group | IV Acetaminophen-Active | IV Vitamin C-Active | Acetaminophen-Placebo | Vitamin C-Placebo
Number analyzed (Participants) | 223 | 40 | 197 | 21
Participants | 58 | 6 | 60 | 9
Statistical Analysis 1: Comparison: IV Acetaminophen-Active vs Acetaminophen-Placebo; Test type: Superiority; p = 0.31, Chi-squared; Risk Difference (RD) = -4.4, 95% CI 2-sided [-13.1 to 4.2]
Statistical Analysis 2: Comparison: IV Vitamin C-Active vs Vitamin C-Placebo; Test type: Superiority; p = 0.02, Chi-squared; Risk Difference (RD) = -27.9, 95% CI 2-sided [-51.7 to -4.0]

17. Secondary Outcome: 90-day Hospital Mortality
Description: Vital status prior to discharge home before day 90.
Time Frame: 90 days after randomization
Measure: Count of Participants; unit: Participants
Arm/Group | IV Acetaminophen-Active | IV Vitamin C-Active | Acetaminophen-Placebo | Vitamin C-Placebo
Number analyzed (Participants) | 224 | 40 | 197 | 21
Participants | 50 | 6 | 45 | 9
Statistical Analysis 1: Comparison: IV Acetaminophen-Active vs Acetaminophen-Placebo; Test type: Superiority; p = 0.90, Chi-squared; Risk Difference (RD) = -0.5, 95% CI 2-sided [-8.5 to 7.5]
Statistical Analysis 2: Comparison: IV Vitamin C-Active vs Vitamin C-Placebo; Test type: Superiority; p = 0.02, Chi-squared; Risk Difference (RD) = -27.9, 95% CI 2-sided [-51.7 to -4.0]

18. Secondary Outcome: Number of Subjects Who Developed ARDS Within 7 Days of Randomization
Description: The presence of ARDS for each day is defined as receiving assisted ventilation with P/F <300 or imputed P/F <300, FiO2 ≥40%, and PEEP ≥5 cm H2O and not fully explained by CHF or fluid overload. ARDS imaging criteria are met if clinically available chest images (CT or CXR) are consistent with ARDS (bilateral opacities not fully explained by effusions, lobar/lung collapse, or nodules).
Time Frame: Up to day 7
Measure: Count of Participants; unit: Participants
Arm/Group | IV Acetaminophen-Active | IV Vitamin C-Active | Acetaminophen-Placebo | Vitamin C-Placebo
Number analyzed (Participants) | 183 | 30 | 169 | 19
Participants | 4 | 2 | 16 | 0
Statistical Analysis 1: Comparison: IV Acetaminophen-Active vs Acetaminophen-Placebo; Test type: Superiority; p = 0.003, Chi-squared; Risk Difference (RD) = -7.3, 95% CI 2-sided [-12.2 to -2.4]
Statistical Analysis 2: Comparison: IV Vitamin C-Active vs Vitamin C-Placebo; Test type: Superiority; p = 0.52, Fisher Exact; Risk Difference (RD) = 6.7, 95% CI 2-sided [-2.3 to 15.6]

19. Secondary Outcome: Change in Serum Creatinine Concentration
Description: We will measure the change in serum creatinine from enrollment to discharge, death, initiation of dialysis or 28 days, whichever occurs first
Time Frame: Up to day 28
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | IV Acetaminophen-Active | IV Vitamin C-Active | Acetaminophen-Placebo | Vitamin C-Placebo
Number analyzed (Participants) | 198 | 37 | 181 | 19
mg/dL | -0.3 (1.0) | -0.2 (1.2) | -0.2 (1.0) | -0.1 (0.3)
Statistical Analysis 1: Comparison: IV Acetaminophen-Active vs Acetaminophen-Placebo; Test type: Superiority; p = 0.68, t-test, 2 sided; Mean Difference (Final Values) = -0.0, 95% CI 2-sided [-0.2 to 0.2]
Statistical Analysis 2: Comparison: IV Vitamin C-Active vs Vitamin C-Placebo; Test type: Superiority; p = 0.62, Fisher Exact; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-0.7 to 0.4]

20. Secondary Outcome: Number of Subjects With Major Adverse Kidney Events at 28 Days (MAKE28)
Description: Defined as persistent increase in serum creatinine by 200% from baseline, need for new renal replacement therapy, or death
Time Frame: 28 days after randomization
Measure: Count of Participants; unit: Participants
Arm/Group | IV Acetaminophen-Active | IV Vitamin C-Active | Acetaminophen-Placebo | Vitamin C-Placebo
Number analyzed (Participants) | 221 | 40 | 197 | 21
Participants | 55 | 9 | 48 | 8
Statistical Analysis 1: Comparison: IV Acetaminophen-Active vs Acetaminophen-Placebo; Test type: Superiority; p = 0.90, Chi-squared; Risk Difference (RD) = 0.5, 95% CI 2-sided [-7.8 to 8.8]
Statistical Analysis 2: Comparison: IV Vitamin C-Active vs Vitamin C-Placebo; Test type: Superiority; p = 0.2, Chi-squared; Risk Difference (RD) = -15.6, 95% CI 2-sided [-40.1 to 8.9]

21. Secondary Outcome: ICU Days to Day 28
Description: ICU free days to day 28 are defined as the number of days spent alive and out of the ICU to day 28.
Time Frame: To day 28
Measure: Mean (Standard Deviation); unit: days
Arm/Group | IV Acetaminophen-Active | IV Vitamin C-Active | Acetaminophen-Placebo | Vitamin C-Placebo
Number analyzed (Participants) | 222 | 40 | 196 | 21
days | 5.3 (6.2) | 6.9 (6.9) | 5.2 (6.2) | 3.8 (6.2)
Statistical Analysis 1: Comparison: IV Acetaminophen-Active vs Acetaminophen-Placebo; Test type: Superiority; p = 0.88, t-test, 2 sided; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-1.1 to 1.3]
Statistical Analysis 2: Comparison: IV Vitamin C-Active vs Vitamin C-Placebo; Test type: Superiority; p = 0.10, t-test, 2 sided; Mean Difference (Final Values) = 3.0, 95% CI 2-sided [-0.6 to 6.6]

ADVERSE EVENTS:
Time Frame: Deaths were assessed up to 90 days post-randomization. Adverse events were assessed up to study day 10 (five days after completion of the study drug infusions) or Hospital discharge, whichever occurs first, with one exception, Major Adverse Kidney Events. Major Adverse Kidney Events (as defined in the protocol) were assessed beyond 10 days for up to 28 days post-randomization. All cause mortality to day 90 for APAP is reported for 223 (4 not reported) and 218 for APAP placebo (2 not reported).
Description: Serious or non-serious events related to study procedures or of uncertain relationship were captured. The number of patients at risk for AEs is all patients randomized to APAP (227) and matching APAP placebo (199; AEs in 19 Vit C shared placebos not included in APAP). For Vit C, number at risk for AEs is all patients randomized to Vit C(40) and matching Vit C placebo (21). Six participants had missing data for the primary outcome and 90 day all cause mortality (2 withdrew consent before day 28).
Arm/Group | IV Acetaminophen-Active | IV Vitamin C-Active | Acetaminophen-Placebo | Vitamin C-Placebo
All-Cause Mortality (participants affected / at risk) | 58/223 | 6/40 | 60/197 | 9/21
Serious Adverse Events (participants affected / at risk) | 20/227 | 4/40 | 18/199 | 4/21
Other Adverse Events (participants affected / at risk) | 12/227 | 2/40 | 7/199 | 2/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IV Acetaminophen-Active (N=227) | IV Vitamin C-Active (N=40) | Acetaminophen-Placebo (N=199) | Vitamin C-Placebo (N=21)
Heart Failure (Nos) (Cardiac disorders) | 1 | 0 | 0 | 0 — Definitely not related
Supraventricular Tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 — Definitely not related
Bowel Obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0 — Probably not related
Ventilator Associated Pneumonia (Infections and infestations) | 1 | 1 | 0 | 0 — Definitely not related
Sepsis (Infections and infestations) | 1 | 0 | 0 | 0 — Definitely not related
AST increased (Investigations) | 2 | 0 | 0 | 0 — Probably not related
Hepatic Function Abnormal (Investigations) | 1 | 0 | 0 | 0 — Probably or possibly related
Function Liver Abnormal (Investigations) | 1 | 0 | 0 | 0 — Definitely not related
Liver Enzyme Abnormal (Investigations) | 2 | 0 | 0 | 0 — Probably or possibly related
Liver Function Tests Multiple Abnormal (Investigations) | 1 | 0 | 0 | 0 — Probably or possibly related
Liver Function Tests Multiple Abnormal (Investigations) | 1 | 0 | 0 | 0 — Probably not related
Myopathy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 — Definitely not related
Embolism Pulmonary (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 — Probably not related
Shock (Vascular disorders) | 1 | 0 | 0 | 0 — Definitely not related
Hypotension (Vascular disorders) | 1 | 0 | 1 | 0 — Probably not related
Hypotension (Vascular disorders) | 1 | 0 | 1 | 0 — Probably or possibly related
Infarct Cerebral (Vascular disorders) | 1 | 0 | 0 | 0 — Definitely not related
Acute Bilateral Popliteal Arterial Occlusion (Vascular disorders) | 1 | 0 | 0 | 0 — Definitely not related
Arrhythmia Ventricular (Cardiac disorders) | 0 | 1 | 0 | 0 — Probably not related
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 — Definitely not related
CVA (Nervous system disorders) | 0 | 1 | 0 | 0 — Definitely not related
Distress Respiratory (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 — Probably not related
Cardiac Arrest (Cardiac disorders) | 0 | 0 | 1 | 0 — Definitely not related
Cardiogenic Shock (Cardiac disorders) | 0 | 0 | 1 | 0 — Definitely not related
Coronary Artery Disease (Cardiac disorders) | 0 | 0 | 1 | 0 — Definitely not related
Cardiomyopathy (Cardiac disorders) | 0 | 0 | 1 | 0 — Definitely not related
Multiple Organ Failure (General disorders) | 0 | 0 | 1 | 0 — Definitely not related
Worsening Infection (Infections and infestations) | 0 | 0 | 1 | 0 — Probably not related
ALT Increased, AST Increased (Investigations) | 0 | 0 | 3 | 0 — Probably not related
AST increased (Investigations) | 0 | 0 | 1 | 0 — Probably or possibly related
Hepatic Function Abnormal (Investigations) | 0 | 0 | 1 | 0 — Definitely not related
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 — Definitely not related
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 — Definitely not related
Thrombosis Venous Deep (Vascular disorders) | 0 | 0 | 1 | 0 — Definitely not related
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0 — Probably not related
Retroperitoneal Hemorrhage Grade 4 (Vascular disorders) | 0 | 0 | 1 | 0 — Definitely not related
Left MCA Stroke (Vascular disorders) | 0 | 0 | 1 | 0 — Probably not related
Ischemic Cardiomyopathy (Cardiac disorders) | 0 | 0 | 0 | 1 — Definitely not related
Atrial Fibrillation Paroxysmal, Tachycardia Ventricular (Cardiac disorders) | 0 | 0 | 0 | 1 — Probably or possibly related
Circulatory Shock (Vascular disorders) | 0 | 0 | 0 | 1 — Definitely not related
Circulatory Shock (Vascular disorders) | 0 | 0 | 0 | 1 — Probably not related
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IV Acetaminophen-Active (N=227) | IV Vitamin C-Active (N=40) | Acetaminophen-Placebo (N=199) | Vitamin C-Placebo (N=21)
Acute Blood Loss Anemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 — Definitely not related
Paroxysmal Atrial Fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0 — Definitely not related
Diabetes Mellitus (Endocrine disorders) | 1 | 0 | 0 | 0 — Probably not related
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 — Definitely not related
Hepatocellular Damage (Hepatobiliary disorders) | 1 | 0 | 0 | 0 — Definitely not related
ALT Increased, AST Increased (Investigations) | 1 | 0 | 0 | 0 — Probably not related
ALT Increased, AST Increased (Investigations) | 1 | 0 | 0 | 0 — Probably or possibly related
Liver Function Tests Multiple Abnormal (Investigations) | 1 | 0 | 0 | 0 — Probably not related
Elevated LFTs (Investigations) | 1 | 0 | 0 | 0 — Probably or possibly related
Hypokalemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 — Probably not related
Kidney Failure Acute (Renal and urinary disorders) | 1 | 0 | 0 | 0 — Definitely not related
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 — Definitely not related
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 — Definitely not related
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 — Probably or possibly related
Transfer Back To ICU (Surgical and medical procedures) | 1 | 0 | 0 | 0 — Definitely not related
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0 — Definitely not related
Pain And Swelling at the Site of Infusion (General disorders) | 0 | 1 | 0 | 0 — Definitely not related
Anemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 — Probably not related
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 0 — Probably or possibly related
Bradycardia (Cardiac disorders) | 0 | 0 | 1 | 0 — Definitely not related
Edema Left Leg (General disorders) | 0 | 0 | 1 | 0 — Definitely not related
Infection Bacterial (Infections and infestations) | 0 | 0 | 1 | 0 — Definitely not related
Hypokalemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 — Definitely not related
Coughing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 — Definitely not related
Fever (General disorders) | 0 | 0 | 0 | 1 — Definitely not related
Headache (Nervous system disorders) | 0 | 0 | 0 | 1 — Probably or possibly related
Altered Mental Status (Nervous system disorders) | 0 | 0 | 0 | 1 — Definitely not related

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (6):
  • Study Protocol: ASTER Protocol version 4.2 (2021-06-08): https://cdn.clinicaltrials.gov/large-docs/08/NCT04291508/Prot_000.pdf
  • Study Protocol: ASTER Protocol version 4.5 (2023-04-25): https://cdn.clinicaltrials.gov/large-docs/08/NCT04291508/Prot_001.pdf
  • Statistical Analysis Plan (2023-09-21): https://cdn.clinicaltrials.gov/large-docs/08/NCT04291508/SAP_002.pdf
  • Informed Consent Form: Stamped-ICD_P1_master_v4 (2021-07-14): https://cdn.clinicaltrials.gov/large-docs/08/NCT04291508/ICF_003.pdf
  • Informed Consent Form: Stamped-ICD_P1_master_v5 (2022-07-27): https://cdn.clinicaltrials.gov/large-docs/08/NCT04291508/ICF_004.pdf
  • Informed Consent Form: ICD_p2_template (2022-07-07): https://cdn.clinicaltrials.gov/large-docs/08/NCT04291508/ICF_007.pdf